CLINICAL TRIAL: NCT04634513
Title: Phase 1 Study of the Safety, Tolerability, and Immunogenicity of Oral Doses of CVD 1208S-122, a Prototype Attenuated Shigella Flexneri 2a Live Vector Expressing Enterotoxigenic Escherichia Coli Antigens
Brief Title: Shigella CVD 31000: Study of Responses With Shigella-ETEC Vaccine Strain CVD 1208S-122
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Wilbur Chen, MD, MS, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00094148
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Shigella Infection; Enterotoxigenic Escherichia Coli Infection
Keywords: vaccine; strain CVD 1208S-122
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Shigella Vaccine at 10^8 cfu or Placebo (Experimental): 3:1 randomization to one dose of vaccine or placebo (Cohort n=8)
  Interventions: Biological: strain CVD 1208S-122; Other: Placebo
- Cohort 2: Shigella Vaccine at 10^9 cfu or Placebo (Experimental): 3:1 randomization to one dose of vaccine or placebo (Cohort n=8)
  Interventions: Biological: strain CVD 1208S-122; Other: Placebo
- Cohort 3: Shigella Vaccine at 10^10 cfu or Placebo (Experimental): 3:1 randomization to one dose of vaccine or placebo (Cohort n=8)
  Interventions: Biological: strain CVD 1208S-122; Other: Placebo
- Cohort 4: Shigella Vaccine or Placebo (Experimental): 2:2:1 randomization to receive either two doses of vaccine, 1 dose of vaccine and one dose of placebo, or two doses of placebo at Days 1 and 29 (Cohort n=30)
  Interventions: Biological: strain CVD 1208S-122; Other: Placebo

INTERVENTIONS:
Biological: strain CVD 1208S-122 — Live, attenuated, vaccine strain of S. flexneri 2a expressing CFA/I and LT of enterotoxigenic E. coli
Other: Placebo — Sodium bicarbonate buffer

SUMMARY:
The purpose of this study is to determine whether a live, oral, combined Shigella-ETEC vaccine candidate, known as strain CVD 1208S-122, is safe and immunogenic.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a live, oral, combined Shigella-ETEC vaccine candidate, known as strain CVD 1208S-122, is safe and immunogenic. This will be a phase 1, double-blind, placebo-controlled, dose-escalating, single-center study, involving three vaccine dosage escalation cohorts (10^8, 10^9, and 10^10 cfu vaccine organisms). Each of the three dose-escalation cohorts will consist of 8 study participants who will be randomly allocated to receive either vaccine (n=6) or placebo (n=2), as a single, oral dose. An independent Safety Monitoring Committee (SMC) will review the available safety data for Cohorts 1 - 3 through 7 days post-vaccination before proceeding to the enrollment of the next cohort. The fourth cohort will be an adaptive design cohort consisting of 30 study participants to be randomly allocated to receive either two doses of vaccine (n=12), one dose of vaccine (n=12), or two doses of placebo (n=6), with the dosage selection based on the highest well-tolerated dose in the dose-escalation cohorts (1 - 3), as determined by the SMC.

Each of the dose-escalation cohorts (1 - 3) will receive the oral dose of blinded study product while in the inpatient setting. During the following subsequent 96 hours (4 days), participants will remain on the inpatient research isolation ward to be closely monitored, and each stool will be collected by study staff. The evaluation and monitoring of participants enrolled in the fourth cohort will be conducted entirely in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 49 years of age
* Written informed consent provided
* Determined to be in good health* based on medical history and review of concomitant medications

  *Good health as defined by an absence of an active chronic medical condition which requires daily prescription medication(s). Participants may be eligible if the medical condition only requires infrequent as needed (PRN) medication and if the investigator determines that the condition does not pose a risk to participant safety or the assessment of reactogenicity and immunogenicity. Any chronic medical condition which does not require a daily prescription medication but might pose a risk to a participant with rapid dehydration (i.e., rapid intravascular volume changes) would be ineligible to participate.
* Documented acceptable results from screening laboratory work (defined in Appendix B), including:

  * Complete blood count (CBC) with differential for total white blood cell count (WBC), absolute neutrophil count (ANC), hemoglobin (Hg), platelet count
  * Creatinine, alanine aminotransferase (ALT), total bilirubin
  * Serum Immunoglobulin A (IgA) level
  * Human immunodeficiency virus (HIV) antibody, Hepatitis B surface antigen (HBsAg), Hepatitis C virus antibody (HCV)
  * HLA-B27 histocompatibility testing
  * Serum Beta human chorionic gonadotropin (β-HCG) test, if the participant is a woman of child-bearing potential
* A passing score (≥70%) on a Comprehension Assessment Tool
* Agrees not to participate in another clinical trial during the study period
* Females of child-bearing potential† agree to use an acceptable form of birth control‡ from enrollment and through at least 4 weeks after vaccination

  †Females of child-bearing potential, defined as having not been sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses, if menopausal.

  ‡Acceptable birth control includes barrier methods such as condoms or diaphragms/cervical cap with spermicide; effective intrauterine devices; NuvaRing®; and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill") or alternatively, monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the study vaccination, abstinence from sexual intercourse with a male partner, or sexual relationships with non-male partners.
* Available for up to a 6-day inpatient stay
* For Participants of Cohorts 1-3 during the time when a U.S. Public Health Emergency for COVID-19 exists, SARS-CoV-2 testing must be performed upon admission to the inpatient ward and must document a negative test result prior to vaccination.

Exclusion Criteria:

* A positive pregnancy test at screening or within 24 h prior to study product dosing
* A female who is breastfeeding
* Poor venous access, as defined by inability to obtain venous blood, for screening labs, after 3 venipuncture attempts
* Abnormal vital signs, defined as:

  * Systolic BP >150 mmHg or Diastolic BP >90 mmHg
  * Resting heart rate >100 bpm
  * Oral temperature ≥38.0°C
* Having received prior vaccines for or have had prior infection with ETEC, LT, cholera, or Shigella, within the past 3 years
* History of diarrhea during travel to a developing country within the past 3 years
* History of chronic gastrointestinal illness, including severe dyspepsia, lactose intolerance, or another significant gastrointestinal tract disease (e.g., irritable bowel syndrome, inflammatory bowel syndrome, gastric ulcer disease)
* Regular use (≥once weekly) of laxatives, anti-diarrheal agents, anti-constipation agents, or antacid therapies
* History of major gastrointestinal surgery (uncomplicated laparoscopic appendectomy or cholecystectomy >1-year prior is permitted)
* Abnormal bowel habits, as defined by <3 stools per week or >2 stools per day in the past 6 months
* Use of systemic antimicrobials§ within the past 2 weeks

  * use of topical (skin), otic, or ophthalmic antibiotics is acceptable, if those doses are not expected to result in significant systemic absorption levels
* Use of oral, parenteral or high-dose inhaled steroids within 30 days
* Use of any medication which might affect immune function# within 30 days

  #examples include anti-cancer drugs, immunomodulating monoclonal antibody therapeutics, and rheumatologic therapies
* Diagnosis of schizophrenia or other major psychiatric disease
* Alcohol or drug abuse within last 5 years
* Presence of immunosuppression, which could be due to active neoplastic disease or a history of any hematologic malignancy (excluding resolved non-melanoma skin cancers), radiation therapy, or primary or secondary immunodeficiencies
* History of allergy to quinolone (e.g., ciprofloxacin) or sulpha drugs (e.g., trimethoprim-sulfamethoxazole)
* Known history of seizure disorder (remote history of a childhood seizure disorder which has completely resolved is acceptable)
* Occupation involving the handling of ETEC, cholera, or Shigella bacteria
* Occupation in food handling industry or care of very young children (<2 years old), elderly (≥70 years), or immunocompromised
* During the time when a U.S. Public Health Emergency for COVID-19 exists, within 14 days prior to the time of vaccination, the presence of 2 or more of any of the following symptoms: fever (≥38°C, chills, myalgia, headache, sore throat, or new olfactory and taste disorder
* During the time when a U.S. Public Health Emergency for COVID-19 exists, within 14 days prior to the time of vaccination, the presence of 1 or more of any of the following respiratory symptoms: cough which cannot otherwise be explained, shortness of breath, or difficulty breathing
* Any other criteria which, in the investigator's opinion, would compromise the safety of the study, the ability of a subject to participate, or the results of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilbur Chen, MD, MS, Principal Investigator — Center for Vaccine Development and Global Health, University of Maryland School of Medicine
Locations (1):
- University of Maryland, Baltimore, University of Maryland School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Cohorts 1-3, individuals received vaccine or placebo, according to random assignment and double-blinded conditions. In Cohort 4, individuals received either 2 doses of vaccine, 1 dose of vaccine, or only placebo; according to random assignment and double-blinded conditions. The reporting of outcomes discriminates those allocated to vaccine vs. placebo.
Groups:
- Cohort 1: Shigella Vaccine at 10^8 Cfu; Cohort 2: Shigella Vaccine at 10^9 Cfu; Cohort 3: Shigella Vaccine at 10^10 Cfu: 3:1 randomization to one dose of vaccine or placebo (Cohort n=8)
  strain CVD 1208S-122: Live, attenuated, vaccine strain of S. flexneri 2a expressing CFA/I and LT of enterotoxigenic E. coli
- Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo: 3:1 randomization to one dose of vaccine or placebo (Cohort n=8)
  Placebo: Sodium bicarbonate buffer
- Cohort 4: Shigella 2-Dose Vaccine; Cohort 4: Shigella 1-Dose Vaccine: 2:2:1 randomization to receive either two doses of vaccine, 1 dose of vaccine and one dose of placebo, or two doses of placebo at Days 1 and 29 (Cohort n=30)
  strain CVD 1208S-122: Live, attenuated, vaccine strain of S. flexneri 2a expressing CFA/I and LT of enterotoxigenic E. coli
- Cohort 4: Placebo: 2:2:1 randomization to receive either two doses of vaccine, 1 dose of vaccine and one dose of placebo, or two doses of placebo at Days 1 and 29 (Cohort n=30)
  Placebo: Sodium bicarbonate buffer
Period: Overall Study
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Started | 6 | 2 | 5 | 2 | 6 | 2 | 12 | 12 | 6
Completed | 6 | 2 | 5 | 2 | 6 | 2 | 12 | 12 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo | Total
Number analyzed (Participants) | 6 | 2 | 5 | 2 | 6 | 2 | 12 | 12 | 6 | 53
Age, Continuous [Mean (Full Range); unit: years] | 31 [23 to 43] | 36.5 [26 to 47] | 31.8 [28 to 37] | 38 [28 to 48] | 29.3 [18 to 44] | 39 [33 to 45] | 32.6 [23 to 42] | 32.7 [20 to 43] | 32.7 [27 to 44] | 32.45 [18 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 1 | 2 | 2 | 6 | 4 | 2 | 21
  Male | 3 | 1 | 5 | 1 | 4 | 0 | 6 | 8 | 4 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 6 | 2 | 5 | 2 | 6 | 1 | 12 | 10 | 6 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 4 | 13
  White | 2 | 2 | 3 | 2 | 5 | 2 | 7 | 9 | 2 | 34
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Fever, Diarrhea, or Dysentery; Solicited Local Adverse Events; Solicited Systemic Adverse Events; and Clinical Safety Laboratory Adverse Events
Description: Participants experiencing fever, diarrhea, or dysentery; solicited local adverse events; solicited systemic adverse events; and clinical safety laboratory adverse events
Time Frame: Solicited AEs: Cohorts 1-3 during 4 days of inpatient and memory aid for another 3 days; Cohort 4 memory aid over 7 days after each dose of study product Clinical Safety Labs: Cohorts 1-3: Day 1 and Day 8; Cohort 4: Days 1 and 29 and Days 8 and 36
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 2 | 5 | 2 | 6 | 2 | 12 | 12 | 6
Participants | 2 | 0 | 2 | 1 | 5 | 0 | 8 | 6 | 3

2. Primary Outcome: Vaccine Organisms Shed in Stools in Cohorts 1-3 - Cohorts 1-3
Description: Vaccine organisms shed in stools in Cohorts 1-3
Time Frame: 7 days
Population: Only cohorts 1-3 are included in this outcome.
Measure: Median (Inter-Quartile Range); unit: CFU/mL
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 2 | 5 | 2 | 6 | 2 | 0 | 0 | 0
CFU/mL | 694500 [239500 to 1500000] | 0 [0 to 0] | 1,130,000 [99000 to 52,100,000] | 0 [0 to 0] | 15,760,000 [6,473,000 to 41,000,000] | 0 [0 to 0] |  |  |

3. Primary Outcome: Vaccine Organisms Shed in Stools in Cohort 4
Description: Vaccine organisms shed in stools in Cohort 4
Time Frame: 2 days
Population: Only cohort 4 was analyzed in this outcome
Measure: Mean (Inter-Quartile Range); unit: CFU/mL
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 6
CFU/mL |  |  |  |  |  |  | 11805 [1733 to 313750] | 1510 [47.75 to 42050] | 0 [0 to 0]

4. Primary Outcome: Number of Participants With Genetically Stable Fecal Shed Organisms
Description: Fecal shed organisms found to be genetically stable, as defined as being PCR positive for Shigella (ipaH or virG), CFA/I (cfaB), and LTB (eltB)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 2 | 5 | 2 | 6 | 2 | 12 | 12 | 6
Participants | 6 | 0 | 5 | 0 | 6 | 0 | 10 | 9 | 0

5. Secondary Outcome: Participants With ELISA Antibody Responses
Description: Seroconversions (defined as 4-fold or higher compared to baseline) in antigen-specific ELISA antibody responses
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 2 | 5 | 2 | 6 | 2 | 12 | 12 | 6
Participants
  LPS IgG | 2 | 0 | 0 | 0 | 6 | 0 | 4 | 2 | 0
  IpaB IgG | 1 | 0 | 1 | 0 | 4 | 0 | 2 | 3 | 0
  CFA/I IgG | 6 | 0 | 4 | 0 | 4 | 0 | 8 | 7 | 0
  LT IgG | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  LPS IgA | 1 | 0 | 3 | 0 | 5 | 0 | 2 | 2 | 0
  IpaB IgA | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0
  CFA/I IgA | 6 | 0 | 3 | 0 | 4 | 0 | 6 | 3 | 0
  LT IgA | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Participants With ASC Responses
Description: Responses (defined as ≥8 spot forming cells/10^6 PBMC) in antigen-specific ASC responses post-vaccination
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
Number analyzed (Participants) | 6 | 2 | 5 | 2 | 6 | 2 | 11 | 11 | 6
Participants
  LPS IgG | 4 | 0 | 2 | 0 | 4 | 0 | 6 | 3 | 0
  IpaB IgG | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 0
  CFA/I IgA | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 0
  LT IgG | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  LPS IgA | 6 | 0 | 3 | 0 | 5 | 0 | 9 | 7 | 0
  IpaB IgA | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 0
  LT IgA | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cohort 1: Shigella Vaccine at 10^8 Cfu | Cohort 1: Placebo | Cohort 2: Shigella Vaccine at 10^9 Cfu | Cohort 2: Placebo | Cohort 3: Shigella Vaccine at 10^10 Cfu | Cohort 3: Placebo | Cohort 4: Shigella 2-Dose Vaccine | Cohort 4: Shigella 1-Dose Vaccine | Cohort 4: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/5 | 0/2 | 0/6 | 0/2 | 0/12 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/5 | 0/2 | 0/6 | 0/2 | 0/12 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 0/2 | 3/5 | 1/2 | 4/6 | 1/2 | 2/12 | 2/12 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Shigella Vaccine at 10^8 Cfu (N=6) | Cohort 1: Placebo (N=2) | Cohort 2: Shigella Vaccine at 10^9 Cfu (N=5) | Cohort 2: Placebo (N=2) | Cohort 3: Shigella Vaccine at 10^10 Cfu (N=6) | Cohort 3: Placebo (N=2) | Cohort 4: Shigella 2-Dose Vaccine (N=12) | Cohort 4: Shigella 1-Dose Vaccine (N=12) | Cohort 4: Placebo (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Streptococcal Sore Throat (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral Syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dog Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wrist Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Absolute Neutrophil Count Decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Bilirubin Total Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Pressure Diastolic Decreased (Investigations) | 2 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Blood Pressure Diastolic Increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Systolic Decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart Rate Decreased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Heart Rate Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Platelet Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Athralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Narcolepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive Urgency (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT04634513/Prot_SAP_000.pdf